CLINICAL TRIAL: NCT05615545
Title: Safety and Efficacy of Cryoablation in the Treatment of Advanced Bone and Soft Tissue Tumors: a Single-center Retrospective Study
Brief Title: Cryoablation for Advanced Bone and Soft Tissue Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Jiaqiang, associate chief physician, Henan Cancer Hospital
Other Study IDs: ZZUSC-10
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-11

CONDITIONS: Sarcoma; Cryoablation
MeSH Terms: conditions — Sarcoma | interventions — Cryosurgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cryoablation: Cryoablation of selected tumor lesions
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Cryoablation — Cryoablation of selected tumor lesions

SUMMARY:
This is a single-center, open, retrospective clinical study of patients with metastatic/surgically unresectable bone and soft tissue sarcoma undergoing cryoablation of selected tumor lesions. All eligible patients were enrolled. Basic data and treatment methods of these patients were collected, and efficacy and safety were evaluated.

DETAILED DESCRIPTION:
This is a single-center, open, retrospective clinical study of patients with metastatic/surgically unresectable bone and soft tissue sarcoma undergoing cryoablation of selected tumor lesions. Clinical data of eligible patients were scheduled to be retrospectively collected from December 2016 to February 28, 2022. All patients eligible for inclusion. Basic data and treatment methods of these patients were collected, and efficacy and safety were evaluated.

ELIGIBILITY:
Inclusion Criteria:

No age restriction, male or female.

The pathological diagnosis was a subtype of bone and soft tissue sarcoma.

The clinical stage was determined to be metastatic or locally unresectable bone and soft tissue sarcoma.

At least one cryoablation of tumor lesions was performed in our hospital.

Target lesions can be evaluated according to the efficacy evaluation criteria for solid tumors (RECIST; Version 1.1) Measure diameter changes.

Follow-up data were complete.

Exclusion Criteria:

Not applicable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cryoablation of selected tumor lesions in patients with metastatic/operatively unresectable bone and soft tissue sarcomas
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-10-28 (Estimated); Study Completion 2024-10-28 (Estimated)

PRIMARY OUTCOMES:
Survival rates | 12 months after surgery
  1-year survival rate
There was no local recurrence survival rate | 12 months after surgery
  The 1-year survival rate without local recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue ,Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No